CLINICAL TRIAL: NCT00163995
Title: Urotensin II and Vascular Tone in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Other Study IDs: AH4004
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2005-09

CONDITIONS: Liver Diseases; Cirrhosis
Keywords: Chronic Liver Disease
MeSH Terms: conditions — Liver Diseases; Fibrosis | interventions — urotensin II

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: urotensin II

SUMMARY:
This study looks at the iontophoresis of urotensin II in chronic liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William W Kemp, MBBS, FRACP, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia